CLINICAL TRIAL: NCT04629040
Title: The Effect of Lateral Wedge Insole for Knee Osteoarthritis Patient in Plantar Pressure, Quadriceps Thickness, Gait and Walking Speed: a Randomized Controlled Trial
Brief Title: The Effect of Lateral Wedge Insole for Knee Osteoarthritis Patient in Plantar Pressure, Quadriceps Thickness, Gait and Walking Speed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH109-REC1-129
Record Dates: First submitted 2020-10-27; First posted 2020-11-16 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Lateral wedge insole
- Control (Placebo Comparator)
  Interventions: Other: Ordinary insole

INTERVENTIONS:
Other: Lateral wedge insole — Lateral wedge insole for knee osteoarthritis patient
  Arms: Intervention
Other: Ordinary insole — Ordinary insole
  Arms: Control

SUMMARY:
Investigators would let knee osteoarthritis patient dressing lateral wedge insole and evaluate the effect for foot pressure modification, quadriceps thickness detected with ultrasound and gait. Investigators would made the patient in control group dressing ordinary insole.

DETAILED DESCRIPTION:
Knee osteoarthritis is one of the most popular disease affected elderly people and made them discomfort. There was no study using foot pressure as a parameter about lateral wedge insole intervention for the knee osteoarthritis patient. The purpose of this study was to investigate the effect of lateral wedge insole for the patient of knee osteoarthritis. During total period of 12 weeks for the study, investigators randomized the patient into experimental and control group. Then investigators evaluated the patient's foot pressure, quadriceps thickness, stride length, stride width, walking speed, pain scale and daily function before intervention, 4th weeks, 8th weeks and 12th weeks. Investigators would use pressure insole designed in the Industrial Technology Research Institute in Taiwan. The portable device used in this study maybe suitable for evaluation of other lower limb disease. There were studies evaluating elderly people dysfunction, critical illness muscle atrophy or knee joint disease with ultrasound detected quadriceps thickness. But there was no study about the correlation between foot pressure and quadriceps thickness for evaluating the effect of lateral wedge insole. Investigators hoped to make a new model for evaluating lower limbs disorder in the future.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis patients
* Medial knee pain

Exclusion Criteria:

* Unable to walk independently
* Ambulation with device
* Any neurologic disease
* Rheumatoid arthritis, gouty arthritis
* History of lower limbs fracture
* History of operation for lower limbs
* Any infectious disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in foot pressure at week 12 | Baseline and week 12
  Investigators would use pressure insole to detect foot pressure of participants at baseline and 12 weeks after dressing insole
Change from baseline in quadriceps thickness at week 4, week 8 and week 12 | Baseline, week 4, week 8 and week 12
  Investigators would use ultrasound to measure quadriceps thickness of participants at baseline, 4 weeks after dressing insole, 8 weeks after dressing insole and 12 weeks after dressing insole

CONTACTS AND LOCATIONS:
Locations (1):
- Asia University Hospital, Taichung, Taiwan